CLINICAL TRIAL: NCT00702442
Title: Role of Droperidol in Postoperative Vomiting: Phase IV Study
Brief Title: Role of Droperidol in Postoperative Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: AHEPA University Hospital (Other)
Responsible Party: Assistant Professor Isaak Kesisoglou, 3rd Department of Surgery, AHEPA University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 597/4-6-2008
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2009-09

CONDITIONS: Vomiting
Keywords: Nausea, Vomiting; Vomiting episodes
MeSH Terms: conditions — Vomiting; Nausea | interventions — Droperidol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): Placebo Administrated 30min prior to operation
  Interventions: Drug: Saline solution
- B (Experimental): 0.625 mg Droperidol administrated i.v 30 min prior surgery
  Interventions: Drug: Droperidol

INTERVENTIONS:
Drug: Droperidol — 0.625 mg droperidol administrated i.v prior to laparoscopic cholecystectomy
  Arms: B
Drug: Saline solution — Saline solution administrated i.v 30 min prior surgery
  Arms: A

SUMMARY:
Protocol title: Role of low dose droperidol in postoperative vomiting

Purpose: Evaluate the efficacy of droperidol to postoperative nausea and vomiting when administrated at the introduction to anesthesia, prior to surgery

Design: Prospective, randomized, placebo-controlled study

Patient Population: Male or female subjects 18 years of age or older who are scheduled for laparoscopic cholecystectomy

No. of Subjects: 100 patients divided into two groups, estimated up to 6 months to enroll

Duration of Treatment: Prior operation

Duration of Follow-up: Follow-up will be performed for 24 hours postoperatively

Endpoints: To evaluate the effectiveness of low dose droperidol when administered Prior surgery

DETAILED DESCRIPTION:
In this prospective, randomized, placebo-controlled study, the researchers determined whether 0.625 mg (1/2 amp) IV droperidol given at the initiation of general anesthesia reduces the incidence of immediate and delayed post operative nausea and vomiting (PONV) in laparoscopic cholecystectomy population. One hundred patients receiving general anesthesia for laparoscopic cholecystectomy received droperidol 0.625 mg (1/2 amp) mg or placebo prior operation.

ELIGIBILITY:
Inclusion Criteria:

* Patient more than 18 years old
* Patients scheduled for laparoscopic cholecystectomy
* Informed consent obtained from the patient

Exclusion Criteria:

* Age < 18 years old
* Contraindication to laparoscopic surgery
* Present a severe depressive syndrome
* Pregnancy women
* Trouble of cardiac rate
* Alcoholism
* Contra-indication for Droperidol prescription

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Vomiting episodes | 24 hours

SECONDARY OUTCOMES:
Light nausea | 24 hours
Control of nausea | 24 hours
Anti-vomiting treatment | 24 hours
Adverse events | 24 hours
Modification of electrocardiograph | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Isaak Kesisoglou, Principal Investigator — Associate Professor in Surgery
Locations (2):
- Greece (2):
  - 3rd Department of Surgery, AHEPA University Hospital, Thessaloniki, Macedonia
  - 3rd Department of Surgery, AHEPA University Hospital, Thessaloniki